CLINICAL TRIAL: NCT04138251
Title: Evaluation of the Safety and Efficacy of Empagliflozin Administration as a Treatment for Neutropenia in Patients With Glycogenosis Type 1b and G6PC3 Deficiency
Brief Title: Safety, Efficacy Evaluation of Empagliflozin Administration for Neutropenia in Glycogenosis Type 1b and G6PC3 Deficiency
Acronym: GLYCO-1B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/26DEC/492
Record Dates: First submitted 2019-06-20; First posted 2019-10-24 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Glycogen Storage Disease Type I; Glucose 6 Phosphatase Deficiency
Keywords: Empaglifozin
MeSH Terms: conditions — Glycogen Storage Disease Type I | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Oral empaglifozin 5 mg 1x/day, increase up to 10 mg 1x/day if no 25% decrease of blood1,5-anhydroglucitol level
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — oral administration of Empagliflozin
  Other Names: Jardiance

SUMMARY:
Treatment of neutropenia of G6PC3 and Glycogenosis type 1b patients with empagliflozin

DETAILED DESCRIPTION:
Ubiquitous glucose-6-phosphatase deficiency (G6PC3) and glucose-6-phosphate transporter deficiency (G6PT/SLC37A4) both cause neutropenia. Studies on a G6PC3 deficient mouse model by Dr Veiga-da-Cunha and Prof. Van Schaftingen and colleagues have shown that these two proteins collaborate to hydrolyze a metabolite that exerts toxic effects on neutrophils. This metabolite is 1,5-anhydroglucitol-6-phosphate. It is formed by phosphorylation of a glucose analogue, 1,5-anhydroglucitol, which is present in the blood of all humans, mice and other mammals.

This discovery of the function of G6PC3 and G6PT opens up therapeutic prospects, in that lowering the concentration of 1,5-anhydroglucitol in the blood should reduce the concentration of 1,5-anhydroglucitol-6-phosphate in the cells and thus reduce its toxic effects. Veiga-da-Cunha, Van Schaftingen and colleagues have already shown that this is the case for a model of mice deficient in G6PC3 treated with empagliflozin .

Following these discoveries, the aim of the investigator's experiment is to test the effect of the efficacy of empagliflozin on urinary excretion and elimination of blood 1,5-anhydroglucitol in patients with glucose-6-phosphate transporter deficiency (type Ib glycogenosis) and patients with G6PC3 deficiency. This should allow patients to significantly lower the level of 1,5-anhydroglucitol-6-phosphate found in their neutrophils and thus cure their neutropenia.

Empagliflozin (marketed in Belgium under the name of Jardiance®) belongs to the class of drugs called oral hypoglycemic agents. It works on the kidney by inhibiting the glucose transporter in the proximal tubules, SGLT2, which leads to glucosuria that results in the elimination of 1,5-anhydroglucitol in the urine. At present, Empagliflozin alone or in combination with other drugs is commonly used in people with type 2 diabetes to control their blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

* Glycogenosis type 1b confirmed by biochemical analyzes and / or genetic analysis. These patients with Glycogenosis must have had a liver transplant
* Alternatively, G6PC3 deficiency confirmed by genetic analysis
* Age 1 to 18 years old female or male
* Informed consent signed by the recipient and / or parents / assigns.
* Information and agreement of the referring medical team.
* A Negative Blood Pregnancy Test at the time of screening and a negative urinary pregnancy test at Day 1 of the protocol are required for female with child bearing potential.
* Sexually active patients should use an effective method of contraception throughout the duration of the study and up to 7 days after the last dose of Empaglifozine. (The combination of a hormonal method and a barrier method; Two barrier methods, the male condom being one of these two methods;Use intrauterine device or tubal ligation;-A total sex abstinence.)

Exclusion Criteria:

* Presence of advanced fibrosis (Metavir F4) or cirrhosis.
* Impossibility of long-term and / or non-compliance monitoring.
* Other medical problems which, in the opinion of the physicians in charge of the patient, would constitute a contraindication to the procedure.
* Sexually active patients who do not consent to use effective contraception during the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Empaglifozin safety (blood test-glycemia): measured by absence of hypoglycaemia due to gliflozin treatment | from start of treatment to 2 months post treatment
  Empaglifozin safety is measured by absence of hypoglycaemia due to gliflozin treatment (continuous monitoring during the first 2 days of treatment and glycemia punctual monitoring every 7 days for 2 months) (mg/dl)
Empaglifozin Efficacy (blood test-hemogram) | from start of treatment to 2 months post treatment
  Efficacy of drug is measured by an Increased neutrophil count as compared to pre-treatment (10exp3/µl)

SECONDARY OUTCOMES:
Empaglifozin Clinical efficacy (questionnaire) | from start of treatment to 2 months post treatment
  Empaglifozin Clinical efficacy is measured as a Decrease in the number of infections
  -Decrease in the number of episodes of oral aphtosis (stomatitis) We will use numerical scale: higher scores mean worse outcome
Empaglifozin Biological efficacy on blood 1,5-anhydroglucitol level (blood test-LCMS) | from start of treatment to 2 months post treatment
  Empaglifozin Biological efficacy is measured as a Decrease of blood 1,5-anhydroglucitol (µM)
Empaglifozin Biological efficacy on 1,5-anhydroglucitol-6-phosphate levels in neutrophils (blood test-LCMS) | from start of treatment to 2 months post treatment
  Empaglifozin Biological efficacy is measured as decrease in the level of 1,5-anhydroglucitol-6-phosphate in neutrophils (µM)
Empaglifozin Clinical efficacy on urinary 1,5-anhydroglucitol excretion increase (urine test-LCMS) | from start of treatment to 2 months post treatment
  Empaglifozin Biological efficacy is measured as increased excretion of urinary 1,5-anhydroglucitol (µM)
Empaglifozin Clinical efficacy on neutrophil function (blood test) | from start of treatment to 2 months post treatment
  Empaglifozin Biological efficacy is measured as improved neutrophilic function (glycosylation analysis, Western Blot)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Stephenne, MD, PhD, Principal Investigator — Cliniques universitaires St Luc
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Proc Natl Acad Sci U S A. 2019 Jan 22;116(4):1241-1250. doi: 10.1073/pnas.1816143116. Epub 2019 Jan 9. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6347702/